CLINICAL TRIAL: NCT03514485
Title: West Philadelphia Asthma Care Implementation Plan
Brief Title: West Philadelphia Controls Asthma
Acronym: WPCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other); Education-Plus, Inc. (Other); The School District of Philadelphia (Other); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 17-013892; 1U01HL138687-01 (NIH)
Record Dates: First submitted 2017-06-26; First posted 2018-05-02 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Childhood Asthma; Community Health Workers
Keywords: asthma disparities; community health worker; childhood asthma
MeSH Terms: interventions — Primary Health Care; Schools

STUDY DESIGN:
Intervention Model Description: A factorial design has enhanced statistical power and can handle cluster randomization of schools. Statistical methods will be used to estimate variation in the effect across schools over time. Linear mixed effects models with random intercepts and slopes for school, and fixed effects for the school-level intervention, time, and time-by-intervention interaction will be applied. Second, marginal models using generalized estimating equations will produce robust estimates that adjust for clustering at the school level. Third, assumption-free, randomization-test-based methods do not rely on assumptions of parametric models. Investigators will use conventional levels of statistical significance (p=0.05) for all pre-specified comparisons for our objectives. Variability of the intervention effect across schools will reflect consistency of intervention effects and thus generalizability in new settings. Both mixed effects models and permutation-test methods will estimate variance components.
Who Masked: Investigator
Masking Description: The Principal Investigator (PI) will be masked to the participant-level intervention group. Unmasking will occur if there is an adverse event that warrants investigation or if the Data Safety and Monitoring Board (DSMB) instructs the PI to become unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- P+S- (Partner School) (Active Comparator): This arm includes children who attend one of the partnering schools and who are randomized to receive the primary care intervention Yes We Can Children's Asthma Program.
  Interventions: Behavioral: Yes We Can Children's Asthma Program
- P-S+ (Partner School) (Active Comparator): This arm includes children who attend one of the partnering schools and who are randomized to receive the school intervention Open Airways for Schools Plus.
  Interventions: Behavioral: Open Airways for School Plus
- P+S+ (Partner School) (Active Comparator): This arm includes children who attend one of the partnering schools and who are randomized to receive the enhanced school intervention Open Airways for Schools Plus, School-Based Asthma Therapy and the primary care intervention Yes We Can Children's Asthma Program.
  Interventions: Behavioral: Yes We Can Children's Asthma Program; Behavioral: School-Based Asthma Therapy; Behavioral: Open Airways for School Plus
- P-S- (Partner School) (No Intervention): This arm includes children who attend one of the partnering schools, and are randomized to the control group (no primary care or school intervention).
- P+ (Non-Partner School) (Active Comparator): This arm includes children who do not attend one of the partnering schools and who are randomized to receive the primary care intervention Yes We Can Children's Asthma Program.
  Interventions: Behavioral: Yes We Can Children's Asthma Program
- P- (Non-Partner School) (No Intervention): This arm includes children who do not attend one of the partnering schools and who are randomized to the control group (no primary care intervention and ineligible for the school intervention).

INTERVENTIONS:
Behavioral: Yes We Can Children's Asthma Program — The Yes We Can Children's Asthma Program intervention is a medical-social model based on a chronic care approach, including risk stratification, clinical care management, social care coordination by a community health worker, and primary care physician asthma champions. This intervention includes asthma education, trigger reduction visits and care coordination. There will be five clinic visits and four home visits over 12 months implemented by the primary care CHW who is integrated into the primary care practice.
  Other Names: Primary Care Intervention
  Arms: P+ (Non-Partner School); P+S+ (Partner School); P+S- (Partner School)
Behavioral: School-Based Asthma Therapy — School-Based Asthma Therapy includes enhanced care coordination for prescribed daily controller medication. The school nurse will coordinate with teachers and the school CHW to schedule daily controller asthma medication administration. The school CHW will assist in obtaining a current asthma care plan and medication administration form from the primary care provider.
  Other Names: Primary Care and School Intervention (Partner School)
  Arms: P+S+ (Partner School)
Behavioral: Open Airways for School Plus — Open Airways for Schools Plus was designed to improve the asthma self-management skills in children and enhance control of asthma in the school. The school intervention includes:
  1. Open Airways for Schools curriculum for all students with asthma. Classes will be conducted by the school CHW once each semester.
  2. Environmental classroom assessments conducted by school CHWs for students enrolled in the study. These teachers will receive classroom supplies to create a more asthma-friendly classroom environment.
  3. Asthma education for school staff/personnel at the start of each school year.
  4. School facility walk-through assessments to detect potential environmental asthma triggers will be conducted by the School District of Philadelphia.
  Other Names: School Intervention (Partner School)
  Arms: P+S+ (Partner School); P-S+ (Partner School)

SUMMARY:
This project uses community health workers (CHW) or lay health educators to implement asthma interventions that have been proven to work in the primary care setting and in schools. The objective is to integrate the home, school, healthcare system, and community for 600 school-aged asthmatic children in West Philadelphia through use of CHWs.

The children enrolled in the study will be randomized to one of four groups including: primary care CHW, school CHW, primary care and school CHW or the control group (no CHW).

DETAILED DESCRIPTION:
The Community Asthma Prevention Program (CAPP) at the Children's Hospital of Philadelphia has a two-decade history of utilizing CHWs to improve asthma outcomes of children in Philadelphia. Building on this foundation, a network of stakeholders was established including, The West Philadelphia Asthma Care Collaborative (WEPACC), with representation from public housing, healthcare, community, and schools. As a result of assessment of local needs, resource mapping, and months of planning, Investigators designed an asthma care implementation program with the broad objective of integrating home, school, healthcare system, and community for school-aged asthmatic children in West Philadelphia. Investigators seek to accomplish this goal using CHWs to deliver sustainable patient-centered evidence-based interventions. The evidence-based interventions include (1) a primary care-based Yes We Can intervention with home visitation and (2) a comprehensive and rigorously evaluated school-based intervention, Open Airways for schools and School Based Asthma Therapy. CHWs will function as the hub of each interventions, serving either as primary care CHWs or school CHWs to provide a network of education, care coordination support, and to facilitate communication for families of children with asthma between the four sectors. This project seeks to integrate interventions in a comprehensive and sustainable manner to reduce asthma disparities in poor, minority children.

Using a factorial design, Investigators will recruit and randomize 640 asthmatic children (ages 5-13 years) from up to five inner-city primary care clinics who attend one of 36 West Philadelphia schools to one of four study conditions: both interventions (both primary care and school CHWs intervention), primary care CHW or school-CHW alone, or control and follow for one year. As a part of this project the Investigators seek to accomplish the following objectives:

Objective 1. Compare effectiveness of the primary care and school interventions to improve asthma control and reduce symptom days using main and simple effects from the factorial design.

Objective 2. Explore moderators and mechanisms of effectiveness and sustainability of the interventions.

Objective 3. Use mixed methods to explore implementation determinants and outcomes of school intervention that promote effectiveness, fidelity and sustainability

Objective 4. Examine the costs, savings, and cost effectiveness associated with the intervention and implementation strategies to promote sustainability.

ELIGIBILITY:
Inclusion Criteria:

1. Children 5-13 years of age and their parents/guardians
2. Children with a diagnosis of asthma
3. Children with uncontrolled asthma (as evidenced within the previous 12 months by an asthma exacerbation requiring oral steroids -OR- an Emergency Department (ED) visit for asthma -OR- an inpatient admission for asthma)
4. West Philadelphia residence in zip code 19104, 19131, 19139, 19142, 19143, 19151 or 19153
5. Children in grades K-8
6. Pediatric primary care received at Children's Hospital of Philadelphia Care Network (CN) Karabots, Cobbs Creek, or South Philadelphia locations or pediatric care received at the Pediatric and Adolescent Medicine Centers of Philadelphia (PAMCOP) serving West Philadelphia residents
7. Parental/guardian permission (informed consent) and, if appropriate, child assent
8. English Language Speaking

Exclusion Criteria:

1. Subjects with other chronic respiratory illnesses such as cystic fibrosis
2. Cyanotic congenital heart disease
3. Mental retardation and/or cerebral palsy (MRCP)
4. Severe Neurological Disorder
5. Cyanotic congenital heart disease
6. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 626 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyra Bryant-Stephens, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Investigators do not plan to share individual level participant data with other researchers, however Investigators plan to make the results (de-identified, aggregate data) available to other researchers and stakeholders interested in asthma and the reduction of asthma disparities. Investigators plan to share results during presentations at organizational and scientific meetings, annual Asthma Summit and published manuscripts. The results will also be shared with the PubMed Data Library.

REFERENCES:
- [Derived] Bryant-Stephens T, Kenyon CC, Tingey C, Apter A, Pappas J, Minto N, Stewart YS, Shults J. Community Health Workers Linking Clinics and Schools and Asthma Control: A Randomized Clinical Trial. JAMA Pediatr. 2024 Dec 1;178(12):1260-1269. doi: 10.1001/jamapediatrics.2024.3967. PMID 39432292

RESULTS

PARTICIPANT FLOW:
Groups:
- P+S+ (Partner School): This arm includes children who attend one of the partnering schools and are randomized to receive the enhanced school intervention Open Airways for Schools Plus, School-Based Asthma Therapy and the primary care intervention Yes We Can Children's Asthma Program.
- P-S+ (Partner School): This arm includes children who attend one of the partnering schools and are randomized to receive the school intervention Open Airways for Schools Plus.
  Open Airways for School Plus: Open Airways for Schools Plus was designed to improve the asthma self-management skills in children and enhance control of asthma in the school. The school intervention includes:
  1. Open Airways for Schools curriculum for all students with asthma. Classes will be conducted by the school community health workers (CHW) once each semester.
  2. Environmental classroom assessments conducted by school CHWs for students enrolled in the study. These teachers will receive classroom supplies to create a more asthma-friendly classroom environment.
  3. Asthma education for school staff/personnel at the start of each school year.
  4. School facility walk-through assessments to detect potential environmental asthma triggers will be conducted by the School District of Philadelphia.
- P+S- (Partner School): This arm includes children who attend one of the partnering schools and are randomized to receive the primary care intervention Yes We Can Children's Asthma Program.
  Yes We Can Children's Asthma Program: The Yes We Can Children's Asthma Program intervention is a medical-social model based on a chronic care approach, including risk stratification, clinical care management, social care coordination by a community health worker, and primary care physician asthma champions. This intervention includes asthma education, trigger reduction visits and care coordination. There will be five clinic visits and four home visits over 12 months implemented by the primary care CHW who is integrated into the primary care practice.
- P-S- (Partner School): This arm includes children who attend one of the partnering schools and are randomized to the control group (no primary care or school intervention).
- P+S0 (Non-Partner School): This arm includes children who do not attend one of the partnering schools and are randomized to receive the primary care intervention Yes We Can Children's Asthma Program.
- P-S0 (Non-Partner School): This arm includes children who do not attend one of the partnering schools and are randomized to the control group (no primary care intervention and ineligible for the school intervention).
Period: Overall Study
Arm/Group | P+S+ (Partner School) | P-S+ (Partner School) | P+S- (Partner School) | P-S- (Partner School) | P+S0 (Non-Partner School) | P-S0 (Non-Partner School)
Started | 121 | 112 | 110 | 112 | 82 | 89
Completed | 116 | 108 | 105 | 111 | 79 | 84
Not Completed | 5 | 4 | 5 | 1 | 3 | 5
Not completed — Lost to Follow-up | 5 | 3 | 2 | 0 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 3 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- P-S+ (Partner School): This arm includes children who attend one of the partnering schools and are randomized to receive the school intervention Open Airways for Schools Plus.
  Open Airways for School Plus: Open Airways for Schools Plus was designed to improve the asthma self-management skills in children and enhance control of asthma in the school. The school intervention includes:
  1. Open Airways for Schools curriculum for all students with asthma. Classes will be conducted by the school CHW once each semester.
  2. Environmental classroom assessments conducted by school CHWs for students enrolled in the study. These teachers will receive classroom supplies to create a more asthma-friendly classroom environment.
  3. Asthma education for school staff/personnel at the start of each school year.
  4. School facility walk-through assessments to detect potential environmental asthma triggers will be conducted by the School District of Philadelphia.
- Total: Total of all reporting groups
Arm/Group | P+S+ (Partner School) | P-S+ (Partner School) | P+S- (Partner School) | P-S- (Partner School) | P+S0 (Non-Partner School) | P-S0 (Non-Partner School) | Total
Number analyzed (Participants) | 121 | 112 | 110 | 112 | 82 | 89 | 626
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 9.3 (2.4) | 8.8 (2.3) | 8.7 (2.6) | 8.4 (2.4) | 8.4 (2.4) | 8.5 (2.4) | 8.7 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 43 | 45 | 40 | 34 | 40 | 263
  Male | 60 | 69 | 65 | 72 | 48 | 49 | 363
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 119 | 103 | 106 | 106 | 79 | 88 | 601
  More than one race | 0 | 5 | 2 | 2 | 2 | 0 | 11
  White | 0 | 1 | 1 | 1 | 0 | 0 | 3
  Asian | 2 | 3 | 1 | 3 | 1 | 1 | 11
BMI [Count of Participants; unit: Participants] — Data reported from Electronic Health Record
  Participants
    < 5th Percentile | 1 | 1 | 0 | 5 | 1 | 2 | 10
    5th to 84th Percentile | 55 | 63 | 45 | 54 | 33 | 42 | 292
    85th to 94th Percentile | 12 | 15 | 15 | 15 | 18 | 12 | 87
    At or Above 95th Percentile | 49 | 31 | 44 | 37 | 28 | 30 | 219
    Missing | 4 | 2 | 6 | 1 | 2 | 3 | 18
Asthma Control Score [Mean (Standard Deviation); unit: units on a scale] — Asthma control was measured using Juniper's Asthma Control Questionnaire (ACQ), a validated instrument with a 6-point scale (with answer values of 0 to 6). The total score is a mean of the 6 answer values. The minimum total score is 0 and the maximum total score is 6. Lower scores indicate better control and a threshold above 1.25 is considered poor control for children. The Minimal Clinically Important Difference (MCID) is 0.5.
  units on a scale | 1.3 (1.3) | 1.4 (1.3) | 1.5 (1.2) | 1.3 (1.2) | 1.3 (1.2) | 1.4 (1.3) | 1.4 (1.3)
Asthma Control Score Groups [Count of Participants; unit: Participants] — Asthma control was measured using Juniper's Asthma Control Questionnaire (ACQ), a validated instrument with a 6-point scale. Lower scores indicate better control and a threshold above 1.25 is considered poor control for children.
  Participants
    0 to <1.25 | 68 | 58 | 51 | 59 | 43 | 49 | 328
    >=1.25 | 52 | 54 | 58 | 53 | 37 | 40 | 294
    Missing | 1 | 0 | 1 | 0 | 2 | 0 | 4
Hospitalized Overnight for Asthma [Count of Participants; unit: Participants] — Data reported from Electronic Health Record
  Participants
    Ever | 78 | 73 | 79 | 71 | 46 | 61 | 408
    Past 12 Months | 36 | 40 | 51 | 33 | 23 | 31 | 214
In the ICU for Asthma [Count of Participants; unit: Participants] — Data reported from Electronic Health Record
  Participants
    Ever | 17 | 12 | 17 | 9 | 9 | 11 | 75
    Past 12 Months | 0 | 1 | 5 | 1 | 1 | 0 | 8
Emergency Department Visit for Asthma [Count of Participants; unit: Participants] — Data reported from Electronic Health Record
  Participants
    Ever | 109 | 94 | 90 | 92 | 74 | 78 | 537
    Past 12 Months | 66 | 60 | 64 | 46 | 43 | 49 | 328
On a Prednisone "Burst" for Asthma [Count of Participants; unit: Participants] — Data reported from Electronic Health Record
  Participants
    Ever | 121 | 112 | 110 | 112 | 82 | 89 | 626
    Past 12 Months | 120 | 112 | 110 | 112 | 82 | 89 | 625
Quality of Life Score (Overall) [Mean (Standard Deviation); unit: units on a scale] — Data was collected using Juniper's Pediatric Asthma Caregiver's Quality of Life Questionnaire designed for children aged 7 to 17 years of age. The PAQLQ has 23 questions in 3 domains (symptoms, activity limitation and emotional function). The activity domain contains 3 'patient-specific' questions within a 1 week recall. The overall score is the mean of all 23 responses and the individual domain scores are the means of the items in those domains. The range is 1-7, with the higher number indicating a better quality of life.
  units on a scale | 5.5 (1.2) | 5.6 (1.2) | 5.2 (1.4) | 5.4 (1.3) | 5.7 (1.1) | 5.5 (1.4) | 5.5 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Asthma Control
Description: Asthma Control Questionnaire (ACQ) developed by E.F. Juniper et al. is a 6-item recall of asthma control indicators over the past week. The 6-item recall includes awakening at night with asthma symptoms, asthma symptoms upon waking, activity limitations due to asthma symptoms, shortness of breath, wheezing, and administration of asthma rescue medications. The score range for the ACQ is 0 to 6, with lower numbers indicating greater asthma control and higher numbers indicating worse asthma control. Based on existing literature, the minimal clinically important difference (MCID) is 0.5. The range for this cohort is 0.2-2.3) For all analyses, we combined the P+S- group with the P+S0 group to describe the P+ only group. Similarly, we combined the P-S- group with the P-S0 group to create the control group.
Time Frame: Baseline and 12 months
Population: P+ Alone group includes children randomized to receive only the primary care intervention. This group combines two arms P+S- and P+S0 (participants who attended a partner school (P+S-) and those who did not attend a partner school (P+S0).
  Similarly, the control group combines P-S- and P-S0 (participants in both groups did not receive any intervention, just usual care).
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- P+S+: This group includes children who attend one of the partnering schools and were randomized to receive both the enhanced school intervention (Open Airways for Schools Plus, School-Based Asthma Therapy) and the primary care intervention (Yes We Can Children's Asthma Program).
- S+ Alone: This group includes children randomized to receive only the enhanced school intervention (Open Airways for Schools Plus, School-Based Asthma Therapy).
- P+ Alone: This group includes children randomized to receive only the primary care intervention (Yes We Can Children's Asthma Program) and combines participants who attended a partner school (P+S-) and those who did not attend a partner school (P+S0).
- Control: This group includes children who were randomized to the control group (no primary care or school intervention) and combines participants who attended a partner school (P-S-) and those who did not attend a partner school (P-S0).
Arm/Group | P+S+ | S+ Alone | P+ Alone | Control
Number analyzed (Participants) | 120 | 112 | 189 | 201
units on a scale
  Baseline | 1.35 [1.16 to 1.54] | 1.42 [1.23 to 1.62] | 1.38 [1.23 to 1.53] | 1.37 [1.22 to 1.51]
  12 Months | 0.74 [0.56 to 0.92] | 0.85 [0.67 to 1.03] | 0.85 [0.72 to 0.99] | 0.97 [0.84 to 1.03]
  Difference (Month 12 minus Baseline) | -0.61 [-0.82 to -0.40] | -0.57 [-0.78 to -0.36] | -0.53 [-0.69 to -0.37] | -0.39 [-0.55 to -0.23]
Statistical Analysis 1: Comparison: P+S+ vs S+ Alone; Linear mixed effects models were then used to make the comparisons of all combinations of primary care and school-based interventions with respect to Asthma Control. Contrasts across time and levels of the intervention were obtained by subtraction. Models were not adjusted for timing of intervention delivery during the Coronavirus (COVID-19) pandemic; Test type: Superiority; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.34 to 0.25]
Statistical Analysis 2: Comparison: P+S+ vs P+ Alone; Linear mixed effects models were then used to make the comparisons of all combinations of primary care and school-based interventions with respect to Asthma Control. Contrasts across time and levels of the intervention were obtained by subtraction. Models were not adjusted for timing of intervention delivery during the COVID-19 pandemic; Test type: Superiority; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.34 to 0.18]
Statistical Analysis 3: Comparison: P+S+ vs Control; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.48 to 0.04]
Statistical Analysis 4: Comparison: S+ Alone vs Control; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.44 to 0.9]
Statistical Analysis 5: Comparison: P+ Alone vs Control; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.36 to 0.09]

2. Secondary Outcome: Change in Daytime Asthma Symptoms
Description: Comparison of the change in daytime symptoms from baseline to 12 months for each intervention group. This data was collected at 3 month intervals with a 2 week recall for number of days with symptoms. This question asks how many days the child has had daytime asthma symptoms in the last 2 weeks and the number of days with asthma symptoms is the answer value (0-14 days).
  P+ Alone group includes children randomized to receive only the primary care intervention. This group combines two arms P+S- and P+S0 (participants who attended a partner school (P+S-) and those who did not attend a partner school (P+S0).
  Similarly, the control group combines P-S- and P-S0 (participants in both groups did not receive any intervention, just usual care).
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: number of symptom days
Arm/Group | P+S+ | S+ Alone | P+ Alone | Control
Number analyzed (Participants) | 118 | 106 | 182 | 194
number of symptom days
  Baseline: number analyzed (Participants) | 118 | 106 | 182 | 193
  Baseline | 1 [0 to 3] | 1.5 [0 to 3] | 1 [0 to 4] | 1 [0 to 3]
  12 Months: number analyzed (Participants) | 117 | 104 | 181 | 194
  12 Months | 0 [0 to 1] | 1 [0 to 2] | 0 [0 to 2] | 1 [0 to 2]
Statistical Analysis 1: Comparison: P+S+ vs S+ Alone; Mixed-effects generalized linear model with binomial family (n=14) was used to make the comparisons of all combinations of primary care and school-based interventions with respect to Daytime Symptoms. Contrasts across time and levels of the intervention were obtained by subtraction. Models were not adjusted for timing of intervention delivery during the Coronavirus (COVID-19) pandemic; Test type: Superiority; Mean Difference (Net) = 0.08, 95% CI 2-sided [-0.39 to 0.55]
Statistical Analysis 2: Comparison: P+S+ vs P+ Alone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.46, 95% CI 2-sided [0.04 to 0.88]
Statistical Analysis 3: Comparison: S+ Alone vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.65, 95% CI 2-sided [-1.06 to -0.23]
Statistical Analysis 4: Comparison: P+ Alone vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Mean Difference (Net) = -1.03, 95% CI 2-sided [-1.39 to -0.67]
Statistical Analysis 5: Comparison: P+S+ vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.57, 95% CI 2-sided [-0.95 to -0.18]

3. Secondary Outcome: Change in Nighttime Symptoms
Description: Comparison of the change in nighttime symptoms from baseline to 12 months for each intervention group. This question asks how many days the child has had nighttime asthma symptoms in the last 2 weeks and the number of days with asthma symptoms is the answer value (0-14 days).
  P+ Alone group includes children randomized to receive only the primary care intervention. This group combines two arms P+S- and P+S0 (participants who attended a partner school (P+S-) and those who did not attend a partner school (P+S0).
  Similarly, the control group combines P-S- and P-S0 (participants in both groups did not receive any intervention, just usual care).
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: number of symptom days
Arm/Group | P+S+ | S+ Alone | P+ Alone | Control
Number analyzed (Participants) | 118 | 107 | 182 | 194
number of symptom days
  Baseline: number analyzed (Participants) | 118 | 107 | 182 | 193
  Baseline | 0 [0 to 2] | 0 [0 to 2] | 0 [0 to 2] | 0 [0 to 2]
  12 Months: number analyzed (Participants) | 116 | 106 | 179 | 194
  12 Months | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 2]
Statistical Analysis 1: Comparison: P+S+ vs S+ Alone; Mixed-effects generalized linear model with binomial family (n=14) was used to make the comparisons of all combinations of primary care and school-based interventions with respect to Nighttime Symptoms. Contrasts across time and levels of the intervention were obtained by subtraction. Models were not adjusted for timing of intervention delivery during the Coronavirus (COVID-19) pandemic; Test type: Superiority; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.53 to 0.28]
Statistical Analysis 2: Comparison: P+S+ vs P+ Alone; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Median Difference (Net) = -0.09, 95% CI 2-sided [-0.45 to 0.26]
Statistical Analysis 3: Comparison: S+ Alone vs Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.25, 95% CI 2-sided [-0.60 to 0.10]
Statistical Analysis 4: Comparison: P+ Alone vs Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Median Difference (Net) = -0.28, 95% CI 2-sided [-0.57 to 0.01]
Statistical Analysis 5: Comparison: P+S+ vs Control; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.38, 95% CI 2-sided [-0.72 to -0.04]

4. Secondary Outcome: Change in School Absences
Description: School report of child's school absences pre and post study enrollment
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | P+S+ | S+ Alone | P+ Alone | Control
Number analyzed (Participants) | 75 | 75 | 61 | 67
days
  Baseline | 11 [3 to 20] | 10 [4 to 23] | 17 [7 to 24] | 13 [7 to 20]
  12 Months | 12 [6 to 26] | 13 [7 to 28] | 16 [7 to 24] | 12 [7 to 23]
Statistical Analysis 1: Comparison: P+S+ vs S+ Alone; Mixed-effects generalized linear model with binomial family (n=number of school-days [varies per child]) was used to make the comparisons of all combinations of primary care and school-based interventions with respect to school absences. Contrasts across time and levels of the intervention were obtained by subtraction. Models were not adjusted for timing of intervention delivery during the Coronavirus (COVID-19) pandemic; Test type: Superiority; Mean Difference (Net) = 2.38, 95% CI 2-sided [0.58 to 4.19]
Statistical Analysis 2: Comparison: P+S+ vs P+ Alone; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; Mean Difference (Net) = 4.49, 95% CI 2-sided [2.54 to 6.43]
Statistical Analysis 3: Comparison: S+ Alone vs Control; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.97, 95% CI 2-sided [-2.78 to 0.84]
Statistical Analysis 4: Comparison: P+ Alone vs Control; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; Mean Difference (Net) = -3.07, 95% CI 2-sided [-5.03 to -1.12]
Statistical Analysis 5: Comparison: P+S+ vs Control; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; Mean Difference (Net) = 1.41, 95% CI 2-sided [-0.48 to 3.31]

5. Secondary Outcome: Change in Emergency Department (ED) Visits
Description: Comparison of the change in asthma-related Emergency Department visits from baseline to 12 months for each intervention group
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: number of ED visits
Arm/Group | P+S+ | S+ Alone | P+ Alone | Control
Number analyzed (Participants) | 121 | 112 | 192 | 201
number of ED visits
  baseline | 1 [0 to 1] | 1 [0 to 2] | 1 [1 to 2] | 1 [0 to 2]
  12 months: number analyzed (Participants) | 118 | 108 | 184 | 198
  12 months | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 1]
Statistical Analysis 1: Comparison: P+S+ vs S+ Alone; Mixed-effects negative binomial models were used to make the comparisons of all combinations of primary care and school-based interventions with respect to number of ED visits. Contrasts across time and levels of the intervention were obtained by subtraction. Models were not adjusted for timing of intervention delivery during the Coronavirus (COVID-19) pandemic; Test type: Superiority; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.19 to 0.54]
Statistical Analysis 2: Comparison: P+S+ vs P+ Alone; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.28 to 0.35]
Statistical Analysis 3: Comparison: S+ Alone vs Control; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.34, 95% CI 2-sided [-0.68 to -0.01]
Statistical Analysis 4: Comparison: P+ Alone vs Control; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.48 to 0.08]
Statistical Analysis 5: Comparison: P+S+ vs Control; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.48 to 0.14]

6. Secondary Outcome: Change in Hospitalizations
Description: Comparison of the change in asthma-related hospitalizations from baseline to 12 months for each intervention group
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: number of hospitalizations
Arm/Group | P+S+ | S+ Alone | P+ Alone | Control
Number analyzed (Participants) | 121 | 112 | 192 | 201
number of hospitalizations
  baseline | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 1]
  12 months: number analyzed (Participants) | 118 | 108 | 184 | 198
  12 months | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: P+S+ vs S+ Alone; Mixed-effects negative binomial models were used to make the comparisons of all combinations of primary care and school-based interventions with respect to number of hospitalizations. Contrasts across time and levels of the intervention were obtained by subtraction. Models were not adjusted for timing of intervention delivery during the Coronavirus (COVID-19) pandemic; Test type: Superiority; Mean Difference (Net) = 0.09, 95% CI 2-sided [-0.11 to 0.29]
Statistical Analysis 2: Comparison: P+S+ vs P+ Alone; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.16, 95% CI 2-sided [-0.03 to 0.34]
Statistical Analysis 3: Comparison: S+ Alone vs Control; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.001, 95% CI 2-sided [-0.19 to 0.18]
Statistical Analysis 4: Comparison: P+ Alone vs Control; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.23 to 0.09]
Statistical Analysis 5: Comparison: P+S+ vs Control; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.09, 95% CI 2-sided [-0.09 to 0.26]

7. Secondary Outcome: Change in Asthma Emotional Functioning Domain
Description: Comparison of the change in caregivers' self-reported quality of life from baseline to 12 months for each intervention group.
  Data was collected using Juniper's Pediatric Asthma Caregiver's Quality of Life Questionnaire designed for children aged 7 to 17 years of age. The PAQLQ has 23 questions in 3 domains, including emotional function. The questions ask about a 1 week recall.
  The range for answer choices is 1-7, with the higher number indicating a better quality of life. The score for the subscale is the mean of the answers for that subscale.
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | P+S+ | S+ Alone | P+ Alone | Control
Number analyzed (Participants) | 120 | 112 | 188 | 199
units on a scale
  Baseline | 5.72 (1.26) | 5.79 (1.18) | 5.55 (1.32) | 5.63 (1.25)
  12 Months: number analyzed (Participants) | 117 | 108 | 182 | 194
  12 Months | 6.47 (0.78) | 6.21 (1.00) | 6.15 (1.08) | 6.16 (1.10)
Statistical Analysis 1: Comparison: P+S+ vs S+ Alone; Mixed-effects linear models with random intercepts for school and child were used to make the comparisons of all combinations of primary care and school-based interventions with respect to QOL emotional functioning domain. Contrasts across time and levels of the intervention were obtained by subtraction. Models were not adjusted for timing of intervention delivery during the Coronavirus (COVID-19) pandemic; Test type: Superiority; Mean Difference (Net) = 0.32, 95% CI 2-sided [0.00 to 0.65]
Statistical Analysis 2: Comparison: P+S+ vs P+ Alone; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.16, 95% CI 2-sided [-0.12 to 0.45]
Statistical Analysis 3: Comparison: S+ Alone vs Control; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.40 to 0.18]
Statistical Analysis 4: Comparison: P+ Alone vs Control; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.20 to 0.29]
Statistical Analysis 5: Comparison: P+S+ vs Control; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.21, 95% CI 2-sided [-0.08 to 0.50]

8. Secondary Outcome: Change in Activity Limitations Domain
Description: Comparison of the change in caregivers' self-reported quality of life from baseline to 12 months for each intervention group.
  he Paediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ) by Juniper et al. is a 13-item measure of asthma caregiver's quality of life in two domains, including activity limitation.
  The score for the subscale is the mean of the answers for the subscale. All items are weighted equally and the score range is 1 - 7, with lower numbers indicating poor quality of life and higher numbers indicating better quality of life around caring for a child with asthma.
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | P+S+ | S+ Alone | P+ Alone | Control
Number analyzed (Participants) | 120 | 112 | 188 | 199
units on a scale
  Baseline | 5.13 (1.51) | 5.18 (1.53) | 5.00 (1.67) | 5.09 (1.69)
  12 Months: number analyzed (Participants) | 117 | 108 | 181 | 194
  12 Months | 6.09 (1.13) | 5.89 (1.25) | 5.79 (1.47) | 5.91 (1.43)
Statistical Analysis 1: Comparison: P+S+ vs S+ Alone; Mixed-effects linear models with random intercepts for school and child were used to make the comparisons of all combinations of primary care and school-based interventions with respect to QOL activity limitations domain. Contrasts across time and levels of the intervention were obtained by subtraction. Models were not adjusted for timing of intervention delivery during the Coronavirus (COVID-19) pandemic; Test type: Superiority; Mean Difference (Net) = 0.25, 95% CI 2-sided [-0.19 to 0.69]
Statistical Analysis 2: Comparison: P+S+ vs P+ Alone; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.25, 95% CI 2-sided [-0.14 to 0.63]
Statistical Analysis 3: Comparison: S+ Alone vs Control; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.49 to 0.30]
Statistical Analysis 4: Comparison: P+ Alone vs Control; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.43 to 0.24]
Statistical Analysis 5: Comparison: P+S+ vs Control; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; Mean Difference (Net) = 0.15, 95% CI 2-sided [-0.24 to 0.54]

9. Secondary Outcome: Baseline School Organizational Climate Index
Description: The Standardized Organizational Climate Index (SOCI) is a 30-item descriptive measure for schools. The index has four dimensions: principal leadership, teacher professionalism, achievement press for students to perform academically, and vulnerability to the community. The score range for each questionnaire item is 1 - 4. The answers assign the value of 1 to "rarely occurs," 2 to "sometimes occurs," 3 to "often occurs," and 4 to "very frequently occurs. For the subscores, ninety-nine percent of the scores range from 200 to 800 with a population mean of 500 and a population standard deviation of 100. Higher scores indicate a better school climate. Scores are converted to standardized scores and compared with national norms.
Time Frame: At start of school intervention
Population: School teachers and staff are the respondents to the surveys, not the children who are the participants of this study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- SOCI Collegial Leadership: SOCI subscale that measures the relationship between principals and teachers.
- SOCI Professional Teacher Behavior: SOCI subscale that captures the relationships among teachers.
- SOCI Achievement Press: SOCI subscale that measures teacher, parental, and principal press for achievement.
- SOCI Institutional Vulnerability: SOCI subscale that evaluates the relationship between the school and community.
Arm/Group | SOCI Collegial Leadership | SOCI Professional Teacher Behavior | SOCI Achievement Press | SOCI Institutional Vulnerability
Number analyzed (Participants) | 253 | 253 | 253 | 253
units on a scale | 538.83 (110.95) | 528.8 (144.88) | 471.46 (121.64) | 441.59 (86.28)

10. Secondary Outcome: Baseline School Leadership
Description: The Implementation Leadership Scale (ILS) is comprised of 12 items assessing the degree to which a leader is Proactive, Knowledgeable, Supportive, and shows Perseverance in implementing evidence-based practice. The range for total score and each subscale score is 0 - 4. Higher scores represent better implementation leadership. The mean of the subscale scores yields the total score.
Time Frame: At start of school intervention
Population: School teachers and staff are the respondents to the surveys, not the children who are the participants of this study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ILS Total: Overall score for Implementation Leadership Scale (ILS), which measures leadership around evidence-based practice implementation.
- ILS Proactive Leadership: Subscale of ILS that refers to the degree to which the leader anticipates and addresses implementation challenges.
- ILS Knowledgeable Leadership: Subscale of ILS that refers to the degree to which a leader has a deep understanding of EBP and implementation issues.
- ILS Supportive Leadership: Subscale of ILS that refers to the leader's support of clinicians' adoption and use of EBP.
- ILS Perseverant Leadership: Subscale of ILS that refers to the degree to which the leader is consistent, unwavering, and responsive to EBP implementation issues.
Arm/Group | ILS Total | ILS Proactive Leadership | ILS Knowledgeable Leadership | ILS Supportive Leadership | ILS Perseverant Leadership
Number analyzed (Participants) | 253 | 253 | 253 | 253 | 253
units on a scale | 1.76 (1.16) | 1.82 (1.24) | 1.57 (1.2) | 1.7 (1.2) | 2.03 (1.27)

11. Secondary Outcome: Baseline School Staff Attitudes
Description: The Evidence-Based Practice Attitude Scale (EBPAS) is a 15-item self-report measure of attitudes toward adoption of EBPs. It consists of four subscales: Appeal (is EBP intuitively appealing), Requirements (would an EBP be used if required), Openness (general openness to innovation), and Divergence (perceived divergence between EBP and current practice). Total score range is 0 - 60. The Appeal, Openness, and Divergence subscales have a range of 0 - 16. The Requirements subscale has a range of 0 - 12. Higher scores indicate more positive attitudes. Subscales are summed to compute a total score.
Time Frame: At start of school intervention
Population: School teachers and staff are the respondents to the surveys, not the children who are the participants of this study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- EBPAS Total: Overall score for attitudes toward evidence-based practices (EBP), in this case asthma interventions in schools.
- EBPAS Requirements: Subscale of EBPAS that refers to the extent to which a staff person will adopt a new practice if required by the organization or legally mandated.
- EBPAS Appeal: Subscale of EBPAS that refers to the extent to which a staff person will adopt a new practice if it is intuitively appealing.
- EBPAS Openness: Subscale of EBPAS that refers to the extent to which a staff person is generally receptive to using new interventions.
- EBPAS Divergence: Subscale of EBPAS that refers the extent to which a staff person perceives research-based treatments as not useful clinically.
Arm/Group | EBPAS Total | EBPAS Requirements | EBPAS Appeal | EBPAS Openness | EBPAS Divergence
Number analyzed (Participants) | 253 | 253 | 253 | 253 | 253
units on a scale | 2.53 (0.65) | 2.31 (1.2) | 2.42 (0.91) | 2.56 (0.87) | 1.01 (0.86)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for up to 12 months.
Arm/Group | P+S+ (Partner School) | P-S+ (Partner School) | P+S- (Partner School) | P-S- (Partner School) | P+S0 (Non-Partner School) | P-S0 (Non-Partner School)
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/112 | 0/110 | 0/112 | 0/82 | 0/89
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/112 | 0/110 | 0/112 | 0/82 | 0/89
Other Adverse Events (participants affected / at risk) | 0/121 | 0/112 | 0/110 | 0/112 | 0/82 | 0/89

LIMITATIONS AND CAVEATS:
This study was conducted during the pandemic. For this reason, the school intervention was disrupted as schools were closed down completely for six months and then only virtual for three months. This prevented us from conducting the school intervention as per protocol for most of the children in the study. This impacted our outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT03514485/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/85/NCT03514485/SAP_001.pdf